CLINICAL TRIAL: NCT00262405
Title: Phase II Trial of Zileuton Compared to Azathioprine/Prednisone for the Treatment of Idiopathic Pulmonary Fibrosis
Brief Title: Zileuton for the Treatment of Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Kevin R. Flaherty, Professor of Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1995-0304; P50HL056402-06 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-12-06 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — zileuton; Azathioprine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- zileuton (Experimental): Zileuton
  Interventions: Drug: zileuton
- azathioprine/prednisone (Active Comparator): azathioprine/prednisone
  Interventions: Drug: azathioprine/prednisone

INTERVENTIONS:
Drug: zileuton
  Arms: zileuton
Drug: azathioprine/prednisone
  Arms: azathioprine/prednisone

SUMMARY:
Open label trial of zileuton compared to azathioprine/prednisone for patients with idiopathic pulmonary fibrosis. Study subjects will undergo a detailed clinical, radiographic, and physiologic assessment at baseline. Subjects will be monitored off treatment for three months for changes in symptoms and physiology. Subjects will then be randomized to six months of treatment with zileuton or azathioprine/prednisone. The primary endpoint of this trial is change in LTB4 levels in bronchoalveolar lavage fluid following six months of treatment. Secondary endpoints are progression free survival, change in dyspnea, change in quality of life, and change in physiology.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic pulmonary fibrosis
* Taking < 15 mg prednisone for at least 30 days prior to screening
* Age 35-80, inclusive
* Able to understand a written informed consent and comply with the study protocol

Exclusion Criteria:

* Significant environmental exposure
* Diagnosis of collagen vascular disease
* Evidence of active infection
* Clinically significant cardiac disease Myocardial infarction, coronary artery bypass or angioplasty within 6mo Unstable angina pectoris Congestive heart failure requiring hospitalization within 6 months Uncontrolled arrhythmia
* Poorly controlled or severe diabetes mellitus
* Pregnancy or lactation
* Women of childbearing potential not using a medically approved means of contraception (i.e. oral contraceptives, intrauterine devices, diaphragm, Norplant)
* Current enrollment in another experimental protocol

Physiologic Criteria:

* FEV1/FVC < 0.60

Laboratory Criteria:

* Total bilirubin > 1.5 X upper limit normal
* AST or ALT > 3X upper limit normal
* Alkaline phosphatase > 3X upper limit normal
* White blood cell count < 2,500/mm3
* Hematocrit < 30%
* Platelets < 100,000/mm3
* Prothrombin time INR > 1.5

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2001-01; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
LTB4 level in BAL | 6 months

SECONDARY OUTCOMES:
CRP score | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Galen B Toews, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States